CLINICAL TRIAL: NCT03330093
Title: Sleep and the Neural Basis of Emotion Processing in Childhood
Brief Title: Sleep and Emotion Processing in Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Monique LeBourgeois, Associate Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0214.04.0421B
Record Dates: First submitted 2017-10-04; First posted 2017-11-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Sleep; Emotions
Keywords: Children
MeSH Terms: interventions — Health

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Extension (Experimental): 1-month educational and problem solving behavioral intervention about sleep.
  Interventions: Behavioral: Sleep Health in Preschoolers
- Health and Safety (Active Comparator): 1-month educational and problem solving behavioral intervention about health and safety.
  Interventions: Behavioral: Health and Safety Intervention

INTERVENTIONS:
Behavioral: Sleep Health in Preschoolers — In-person, family-based behavioral intervention
  Arms: Sleep Extension
Behavioral: Health and Safety Intervention — In-person, family-based behavioral intervention
  Arms: Health and Safety

SUMMARY:
This research project will examine whether experimental sleep extension in children alters the neural and behavioral mechanisms by which short sleep is a risk factor for emotional/behavioral problems. Children ages 5.0-5.9 years with chronic insufficient sleep (≤9 h/night for ≥6 months) will be randomized to either a sleep Extension or to an active Control group. Extension group parents will participate in a 1-month individualized behavioral sleep intervention to promote targeted sleep duration improvements before beginning a 2-week sleep Extension schedule (8 week protocol). Brain and behavioral assessments will occur at Baseline and post sleep Extension.

DETAILED DESCRIPTION:
Research on processes influencing the development of affective brain circuits is critical to elucidating the neurobiological substrates of psychiatric disorders. Mechanistic evidence from adults showing a sleep-dependent functional "disconnect" between brain regions central to adaptive emotion processing (i.e., regulation and expression) suggests that sleep loss is a fundamental target. Similar data in young children, however, do not exist. Early childhood is a sensitive period in the maturation of sleep and emotion processing and also a time when disturbance in both domains is commonly first detected. Further, epidemiological findings reveal that insufficient sleep in childhood is prevalent, associated with concurrent emotional problems, and predicts later mood and attentional disorders. Although the investigator's recent experimental findings indicate that acute sleep loss results in non-adaptive emotion processing in young children, the neural systems underlying such sleep-dependent effects are not known. Also, the vast majority of basic research on sleep and affective substrates has utilized sleep deprivation or sleep restriction protocols. The investigators will instead employ sleep extension in chronically sleep-restricted children, a highly translatable approach with significant public health implications.

This research project will examine whether experimental sleep extension in children alters the neural and behavioral mechanisms by which short sleep is a risk factor for emotional/behavioral problems. Children ages 5.0-5.9 years with chronic insufficient sleep (≤9 h/night for ≥6 months) will be randomized to either a sleep Extension or to an active Control group. Extension group parents will participate in a 1-month individualized behavioral sleep intervention to promote targeted sleep duration improvements before beginning a 2-week sleep Extension schedule (8 week protocol). Brain and behavioral assessments will occur at Baseline and post sleep Extension.

ELIGIBILITY:
Inclusion Criteria:

4.0-6.9 years Reportedly obtain ≤9 h of sleep/night for ≥6 months

Exclusion Criteria:

Nocturnal sleep disturbance determined by clinical cut-offs on the Children's Sleep Habits Questionnaire and the Pediatric Sleep Questionnaire Medications Developmental disabilities Chronic medical conditions Low-birth weight or pre-term term delivery Family history of psychiatric disorders Living at altitude <1 year Metal implants or Claustrophobia

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
MRI/fMRI | Change from Baseline at 10 weeks
  Brain Scans to assess neural substrates of emotion

SECONDARY OUTCOMES:
Emotion Regulation Checklist | Change from Baseline at 10 weeks
  Parent report questionnaire to assess emotion regulation

IPD SHARING:
Plan to Share IPD: No